CLINICAL TRIAL: NCT01281670
Title: The Effects of Combining Whole Body Vibration Training With Plyometric Jumping on the Neuromuscular Adaptations of Human Triceps Surae Muscles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hsing-Kuo Wang/Associate Professor, Natioal Tiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 201009070R
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Muscle Force, Explosive Strength and Vertical Jump Height
Keywords: H reflex; muscle activation; rate of force development; whole body vibration
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No vibration (No Intervention)
- vibration (Active Comparator)
  Interventions: Other: vibration

INTERVENTIONS:
Other: vibration — 8 week vibration
  Arms: vibration

SUMMARY:
Muscle force, explosive strength and vertical jump height are important parameters determining the performance of athletes. Traditionally, high intensity resistance training, explosive strength training and plyometric training are used to improve athletes' performance. Recently, whole body vibration training is recommended for increasing muscle force and explosive strength, because vibrating platform could provide high gravitational acceleration to activate muscle activation and sensory input to spinal reflex. Design: Prospective and randomized control study. Subjects: Healthy male subjects with regular training or competition at least 6 hours per week. Methods: H-reflex, V-wave, triceps surae activation level and rate of force development are measured at pre-training, mid-training (5th week) and post-training. Subjects will receive 8 weeks, 3 times/week, training programs including plyometric jumping or static squat on whole body vibration platform. Data analysis: Data will be analyzed using SPSS 13.0 software (SPSS Inc., Chicago, IL) and two-way ANOVA will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* subjects who had not been engaged in systematic strength training and had no history of knee, leg, or ankle pain that caused a subject to seek medical help during the year prior to the recruitment.

Exclusion Criteria:

* Subjects who missed more than one training session or participated in any other type of fitness training were excluded.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
evoked spinal reflex | 8 weeks
  In terms of evoked spinal reflexes, modulations of spinal inhibitory inter-neuronal circuits are often assessed by the Ia-afferent-mediated H-reflex. Results of H reflexes in studies with training are tightly coupled with excitability changes of small alpha motor neurons. The first volitional (V) wave, an electrophysiological variant of the H-reflex, is used to indicate the net excitation of the motorneurone pool.

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Kuo Wang, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University, Taipei, Taiwan, Taiwan